CLINICAL TRIAL: NCT04408651
Title: Low Intensity Internet Therapy for Chronic Illness (@LIIT.CI): Testing the Efficacy of ACT and CFT Interventions
Brief Title: Low Intensity Internet Therapy for Chronic Illness (@LIIT.CI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Inês A Trindade, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIIT
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Medical Conditions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental)
  Interventions: Behavioral: LIIT.CI ACT
- Compassion-Focused Therapy (Experimental)
  Interventions: Behavioral: LIIT.CI CFT

INTERVENTIONS:
Behavioral: LIIT.CI ACT — 4-week online self-management intervention based on Acceptance and Commitment Therapy and adapted to people with chronic medical conditions
  Arms: Acceptance and Commitment Therapy
Behavioral: LIIT.CI CFT — 4-week online self-management intervention based on Compassion-Focused Therapy and adapted to people with chronic medical conditions
  Arms: Compassion-Focused Therapy

SUMMARY:
Chronic illness (CI) presents a significant and negative effect on quality of life and mental health. Further, emotion regulation has been considered of particular importance on the determination of chronic patients' well-being. Evidence suggests that Acceptance and Commitment Therapy (ACT) is an effective approach to improve psychological health in patients with CI. Further, there is some, although limited, evidence, that self-compassion training may be also useful in this context, and the inclusion of self-compassion elements in ACT interventions has even been the focus of attention by recent studies. Nevertheless, no study yet has compared the efficacy of these two types of intervention in CI. This is the aim of the present project - to analyse, in a low intensity eHealth intervention context, whether ACT or Compassion Focused Therapy (CFT) present superiority over the other in improving mental health and illness-related outcomes in CI.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Previous diagnosis of a physical chronic medical condition
* Easy access to internet and to a computer

Exclusion Criteria:

* Receiving psychological intervention
* Diagnosis of a severe psychiatric disorder (e.g., schizophrenia, bipolar disorder) or cognitive impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Depression and anxiety (Hospital Anxiety and Depression Scales; HADS) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate more depression and anxiety symptoms (0-21)

SECONDARY OUTCOMES:
Illness shame (Chronic Illness Shame Scale; CISS) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate higher levels of illness shame (0-28)
Psychological Flexibility (Comprehensive assessment of ACT processes; CompACT) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate higher levels of psychological flexibility (0-108)
Self-compassion (Self-compassion scale; SCS) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate higher levels of self-compassion (subscale of the Self-compassion scale) (13-65)
Self-criticism (Self-compassion scale; SCS) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate higher levels of self-cristicism (subscale of the Self-compassion scale) (13-65)
Cognitive fusion (Cognitive Fusion Scale; CFQ-7) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate higher levels of cognitive fusion (0-28)

OTHER OUTCOMES:
Fear of contracting COVID-19 (Fear of contracting COVID-19 scale; FCCS) | Changes in results from: immediately pre-intervention and immediately post-intervention assessments
  Higher scores indicate more fear of contracting COVID-19 (9-45)

CONTACTS AND LOCATIONS:
Locations (1):
- Inês Trindade, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided